CLINICAL TRIAL: NCT05981391
Title: An Evaluation of Neurobiological Similarities of Tinnitus and Posttraumatic Stress Disorder
Brief Title: Neurobiological Similarities of Tinnitus and PTSD
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Hearing Center of Excellence (U.S. Federal Agency); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, John Moring, Assistant Professor, The University of Texas Health Science Center at San Antonio
Other Study IDs: HSC20200573HU; 5K23MH122579 (NIH)
Record Dates: First submitted 2023-07-31; First posted 2023-08-08 (Actual); Results first posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Posttraumatic Stress Disorder; Tinnitus
Keywords: resting-state fMRI; PTSD; tinnitus; military; veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Tinnitus | interventions — Acoustic Impedance Tests; Otoscopy; Bone Conduction; Hearing Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Tinnitus and PTSD (T+P): Active duty service members and/or veterans with PTSD and tinnitus.
  Interventions: Diagnostic Test: resting-state functional MRI; Diagnostic Test: Clinician Administered PTSD Scale for the DSM-5 (CAPS-5); Diagnostic Test: Tympanometry; Diagnostic Test: Tinnitus Assessment; Diagnostic Test: Otoscopy; Diagnostic Test: Pure tone air and bone-conduction; Diagnostic Test: Speech testing; Diagnostic Test: Loudness Discomfort; Diagnostic Test: Quick Speech in Noise Test; Diagnostic Test: Distortion-Product Otoacoustic Emissions (DPOAE)
- Tinnitus Only (TO): Active duty service members and/or veterans with only tinnitus/no PTSD.
  Interventions: Diagnostic Test: resting-state functional MRI; Diagnostic Test: Tympanometry; Diagnostic Test: Tinnitus Assessment; Diagnostic Test: Otoscopy; Diagnostic Test: Pure tone air and bone-conduction; Diagnostic Test: Speech testing; Diagnostic Test: Loudness Discomfort; Diagnostic Test: Quick Speech in Noise Test; Diagnostic Test: Distortion-Product Otoacoustic Emissions (DPOAE)
- PTSD Only (PO): Active duty service members and/or veterans with only PTSD/no tinnitus.
  Interventions: Diagnostic Test: resting-state functional MRI; Diagnostic Test: Clinician Administered PTSD Scale for the DSM-5 (CAPS-5); Diagnostic Test: Tympanometry; Diagnostic Test: Otoscopy; Diagnostic Test: Pure tone air and bone-conduction; Diagnostic Test: Speech testing; Diagnostic Test: Loudness Discomfort; Diagnostic Test: Quick Speech in Noise Test; Diagnostic Test: Distortion-Product Otoacoustic Emissions (DPOAE)
- Healthy Controls: Active duty service members and/or veterans with no PTSD and no tinnitus.
  Interventions: Diagnostic Test: resting-state functional MRI; Diagnostic Test: Tympanometry; Diagnostic Test: Otoscopy; Diagnostic Test: Pure tone air and bone-conduction; Diagnostic Test: Speech testing; Diagnostic Test: Loudness Discomfort; Diagnostic Test: Quick Speech in Noise Test; Diagnostic Test: Distortion-Product Otoacoustic Emissions (DPOAE)

INTERVENTIONS:
Diagnostic Test: resting-state functional MRI — We will acquire BOLD fMRI images in an unstimulated state using an extended time-series (300 whole-brain volumes over ~ 60-75 min). These data are a main outcome. Data will be processed on an ongoing basis to ensure integrity, and includes controlling for white matter, cerebral spinal fluid, and movement.
Diagnostic Test: Clinician Administered PTSD Scale for the DSM-5 (CAPS-5) — The CAPS-5 is a semi-structured interview, conducted by an independent evaluator, that measures DSM-5 symptoms of PTSD. Presence of at least one intrusion symptom, one avoidance symptom, two cognition and mood symptoms, and two arousal symptoms for 1 month or more are required to reach the diagnostic threshold.
  Groups: PTSD Only (PO); Tinnitus and PTSD (T+P)
Diagnostic Test: Tympanometry — Tympanometry will be conducted to assess ear canal volume (cm cubed), maximum pressure (daPa) peak compliance (ml), and type (A, AD, AS, B, B-High, C) for each ear) at 226-Hz admittance.
Diagnostic Test: Tinnitus Assessment — Tinnitus acoustic assessment (for tinnitus participants only): Tinnitus ear (left, right, bilateral), pitch matched frequency (Hz) and loudness matched intensity (dB) will be conducted. When available, the tinnitus acoustic assessment only will be repeated at the RII, on the same day and prior to the fMRI scan, to demonstrate reproducibility of results.
  Groups: Tinnitus Only (TO); Tinnitus and PTSD (T+P)
Diagnostic Test: Otoscopy — Otoscopy is a clinical procedure used to examine structures of the ear, particularly the external auditory canal, tympanic membrane, and middle ear
Diagnostic Test: Pure tone air and bone-conduction — Pure tone air- and bone-conduction threshold will be conducted to evaluate audiometry and masking levels in both ears, from 250 Hz. To 16000 Hz.
Diagnostic Test: Speech testing — Speech testing will be conducted in both ears, which will include speech reception threshold, speech reception threshold masking level, word recognition presentation level, and word recognition masking level.
Diagnostic Test: Loudness Discomfort — Loudness discomfort levels will be tested in both right and left ears, from 500Hz to 4000Hz and speech reception threshold.
Diagnostic Test: Quick Speech in Noise Test — Quick Speech in Noise Test (QuickSIN) is a quick method for clinicians to quantify a patient's ability to hear in noise (1 minute).
Diagnostic Test: Distortion-Product Otoacoustic Emissions (DPOAE) — Distortion-Product Otoacoustic Emissions (DPOAE) is an automated evaluation of cochlear function. A sensitive microphone is placed in the ear canal via a probe assembly with a disposable ear-tip attached to perform and record the measurements. DPOAEs will be elicited at multiple frequencies in both ears (10 min).

SUMMARY:
Psychiatric distress caused by PTSD may increase attention toward tinnitus, as well as perceived loudness and discomfort. It is important to understand how tinnitus-related distress and PTSD negatively interact together, in order to develop more effective therapeutic approaches. Understanding symptoms and neurobiological mechanisms using functional magnetic resonance imaging (fMRI), can lead to the necessary knowledge to develop effective interventions for individuals who suffer from both conditions.

DETAILED DESCRIPTION:
Tinnitus and posttraumatic stress disorder (PTSD) are two of the most common service-connected disabilities for active-duty Service Members and Veterans. Tinnitus and PTSD are highly co-morbid, yet distinct disorders. Tinnitus is an auditory disorder in which an illusory auditory percept is experienced, usually as ringing, buzzing, or whooshing sounds, despite no external objective noise source. On the other hand, PTSD is a trauma-related disorder, and is identified by intrusions of the traumatic event, avoidance of reminders, negative alterations in cognition and mood, and hypervigilance or hyperarousal. Similarities between tinnitus and PTSD have been documented among Cambodian refugees, as well as among U.S. Veteran samples. Moreover, the latest neuroimaging data from a recent clinical trial indicated that the auditory-vigilance network was the most dysregulated among active-duty service members with PTSD, compared to combat controls and civilian controls. Due to similar symptoms between tinnitus-related distress and PTSD, and similar dysregulated resting-state brain networks, it remains important to more fully understand how these two distinct disorders may be related. This study will be the first to prospectively examine the overt emotional, behavioral, and cognitive symptoms related to tinnitus-related distress and PTSD, and the overlapping functional connectivity between tinnitus and PTSD. Investigators will examine the overlapping symptoms and neurobiological mechanisms by conducting audiometric and psychological assessments and resting-state functional magnetic resonance imaging (fMRI) among 120 participants (30 with tinnitus and PTSD, 30 with only PTSD, 30 with only tinnitus, and 30 healthy controls). Participants will be recruited from the Frank Tejeda PTSD Clinic and the Audiology Clinic within the South Texas VA Health Care System, and the Hearing Center of Excellence at Lackland Air Force Base. Canonical correlations will be conducted to examine the symptom overlap between tinnitus and PTSD (Aim 1). Investigators aim to neurobiologically characterize tinnitus and PTSD, both separately and conjointly, by conducting fMRI (Aim 2). Investigators also aim to apply modeling to psychometric and neurofunctional data to identify specific regions of the auditory-vigilance network associated with distress related to tinnitus and PTSD. Understanding the shared cognitive, emotional, and behavioral symptoms and neurobiology associated with tinnitus and PTSD will help clinicians and researchers fully understand tinnitus and PTSD independently and conjointly. Results will lead to the identification of neurobiological markers for tinnitus and PTSD, identification of a different phenotype for individuals with both conditions, and development of behavioral and neuro-modulatory therapies that can reduce distress and impairment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female DEERS eligible veterans and active duty service members, ages 18 and above
* preferred language is English and able to read and speak English at a 6th grade level
* those with PTSD (T&P; PO) must meet full criteria for PTSD diagnosis based on the DSM-5 and assessed by an independent evaluator using the CAPS-5
* those with chronic, constant tinnitus (T&P, TO) will be identified by self-report and confirmed with the audiometric assessment.

Exclusion Criteria:

* psychiatric hospitalization in the last 12 months
* significant cognitive impairment determined by inability to comprehend screening assessment
* psychiatric problems and/or high suicide risk warranting immediate intervention
* neurobiological disorders, Meniere's disease
* Temporomandibular disorders that affect tinnitus, per self-report
* history of major head trauma with loss of consciousness for 20 minutes or more as determined by the History of Head Injuries questionnaire
* history of seizures
* conditions that would prevent completion of fMRI scan (any type of electronic, mechanical, or magnetic implant, coil, filter, or stent, any type of surgical clip or staple, shunt, any type of metal object, hearing aid, spinal fusion, halo vest, IV access port, eyelid spring, artificial eye, artificial heart valve, biostimulator, severe hyperacusis)
* active conductive pathology/hearing loss as determined by audiometric assessment.
* Those with tinnitus (T&P; TO) will be excluded if their tinnitus is intermittent, objective, or pulsatile, or present for less than 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will consent and screen veterans and active duty service members to include 120 for analysis. Subjects will be recruited from the San Antonio community. Women and minorities will be actively recruited into the study.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UT Health San Antonio, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tinnitus and PTSD (T+P) | Tinnitus Only (TO) | PTSD Only (PO) | Healthy Controls
Started | 16 | 25 | 3 | 20
Completed | 12 | 24 | 3 | 19
Not Completed | 4 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tinnitus and PTSD (T+P) | Tinnitus Only (TO) | PTSD Only (PO) | Healthy Controls | Total
Number analyzed (Participants) | 16 | 25 | 3 | 20 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.98 (15.28) | 49.39 (15.50) | 47.69 (14.87) | 45.37 (16.00) | 48.89 (15.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 8 | 2 | 7 | 19
  Male | 14 | 17 | 1 | 13 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 1 | 3 | 14
  Not Hispanic or Latino | 13 | 18 | 1 | 17 | 49
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 0 | 5 | 9
  White | 14 | 21 | 1 | 14 | 50
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 16 | 25 | 3 | 20 | 64

OUTCOME MEASURES:

1. Primary Outcome: Resting-State Functional MRI
Description: We will acquire BOLD fMRI images in an unstimulated state using an extended time-series (300 whole-brain volumes over ~ 30 min) and assess for activation within the Auditory Vigilance Network. These data are a main outcome. Data were be processed on an ongoing basis to ensure integrity, and includes controlling for white matter, cerebral spinal fluid, and movement.
  BOLD levels were transformed to Z-scores, a statistical measure that conveys how many standard deviations the data points are away from the dataset. A Z-score of 0 represents the population mean. For each of the regions reported in the Auditory Vigilance Network, each positive point represents one standard deviation above the population mean. These positive Z-scores represent more brain activation within these regions.
Time Frame: 30 minutes of acquired data
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | Tinnitus and PTSD (T+P) | Tinnitus Only (TO) | PTSD Only (PO) | Healthy Controls
Number analyzed (Participants) | 12 | 24 | 3 | 19
Z-Score
  Right Precuneus | 0.55 (0.33) | 0.35 (0.24) | 0.29 (0.22) | 0.59 (0.28)
  Left Cerebellum | 0.46 (0.18) | 0.36 (0.20) | 0.47 (0.27) | 0.54 (0.28)
  Left Superior Temporal Gyrus | 1.80 (0.49) | 1.67 (0.44) | 1.68 (0.45) | 1.95 (0.38)
  Left Cingulate Gyrus | 1.54 (0.47) | 1.60 (0.49) | 1.49 (0.44) | 1.99 (0.38)
  Right Lentiform Nucleus | 1.03 (0.17) | 1.07 (0.19) | 0.97 (0.02) | 1.22 (0.23)
  Right Middle Frontal Gyrus | 0.39 (0.44) | 0.55 (0.32) | 0.37 (0.55) | 0.84 (0.29)
  Left Claustrum | 0.66 (0.20) | 0.73 (0.17) | 0.84 (0.15) | 0.82 (0.26)
  Right Supramarginal Gyrus | 0.53 (0.40) | 0.98 (0.52) | 1.16 (0.97) | 0.95 (0.49)
  Left Insula | 0.24 (0.17) | 0.43 (0.24) | 0.29 (0.11) | 0.40 (0.17)
  Left Medial Frontal Gyrus | 1.32 (0.33) | 0.85 (0.29) | 0.64 (0.08) | 0.96 (0.33)
  Right Insula | 2.32 (0.32) | 2.82 (0.59) | 0.64 (0.48) | 2.86 (0.79)
Statistical Analysis 1: Comparison: Tinnitus and PTSD (T+P) vs Tinnitus Only (TO) vs PTSD Only (PO) vs Healthy Controls; Test type: Superiority; p = 0.01, t-test, 2 sided — Adjusted for multiple comparisons

ADVERSE EVENTS:
Time Frame: 2 months
Description: AEs were assessed each visit. AEs were recorded no matter whether the AE was related to the study.
Groups:
- Healthy Controls: Active duty service members and/or veterans without PTSD and without tinnitus.
Arm/Group | Tinnitus and PTSD (T+P) | Tinnitus Only (TO) | PTSD Only (PO) | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/25 | 0/3 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/25 | 0/3 | 0/24
Other Adverse Events (participants affected / at risk) | 4/12 | 1/25 | 2/3 | 0/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tinnitus and PTSD (T+P) (N=12) | Tinnitus Only (TO) (N=25) | PTSD Only (PO) (N=3) | Healthy Controls (N=24)
Increased PTSD symptoms after evaluation (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
pain from shoulder injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — pain from popped out shoulder during bowling
increased trauma trigger (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — due to break-in at home
increased perceived loudness of tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — due to focus on ringing after entering study
increased tinnitus loudness in both ears (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — after audiometric assessment "maybe psychosomatic"
anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — due to MRI scan

LIMITATIONS AND CAVEATS:
The planned recruitment included 30 participants with both tinnitus and PTSD (T+P); 30 participants with only PTSD (PO); 30 participants with only tinnitus (TO); and 30 healthy controls without PTSD or tinnitus (HC). Groups that were more highly represented included TO (n = 25) and HC (n = 24). Therefore, it is difficult to gain statistical power to assess whether there were significant differences in the BOLD signal for this group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-23): https://cdn.clinicaltrials.gov/large-docs/91/NCT05981391/Prot_SAP_001.pdf
  • Informed Consent Form (2024-04-29): https://cdn.clinicaltrials.gov/large-docs/91/NCT05981391/ICF_000.pdf